CLINICAL TRIAL: NCT02878616
Title: Open-label, Parallel-group, Drug-drug Interaction Study in End-stage Renal Disease Patients Awaiting Kidney Transplant to Investigate the Potential Effect of IVIG Treatment on the Pharmacokinetics and Pharmacodynamics of LFG316
Brief Title: Study in End-stage Renal Disease Patients Awaiting Kidney Transplant to Investigate the Potential Effect of IVIG Treatment on the Pharmacokinetics and Pharmacodynamics of LFG316
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLFG316B2101
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2018-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LFG316 + IVIG (Experimental)
  Interventions: Drug: LFG316; Drug: IVIG
- LFG316 alone (Experimental)
  Interventions: Drug: LFG316

INTERVENTIONS:
Drug: LFG316 — LFG316 single dose
Drug: IVIG — IVIG single dose
  Arms: LFG316 + IVIG

SUMMARY:
Investigate whether concomitant treatment with intravenous immunoglobulin (IVIG) can alter the pharmacokinetics and pharmacodynamics of LFG316 to an extent which would necessitate dose adaptation for LFG316 in pre-sensitized end-stage renal disease patients awaiting kidney transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women 18-70 years of age suffering from end-stage renal disease and who are on chronic dialysis therapy.
2. Candidates for kidney transplantation who are pre-sensitized and will be undergoing desensitization therapy.
3. Written informed consent must be obtained before any assessment is performed.
4. Able to communicate well with the investigator, to understand and comply with the requirements of the study.
5. Recipients who are ABO compatible with donor allograft.
6. Patients awaiting kidney allograft from a living or deceased donor. For patients awaiting transplant from a living donor, kidney transplantation must only occur after 28 days post-LFG316 infusion.
7. History of vaccination with meningococcus and pneumococcus between 2 weeks and 36 months prior to dosing. Documentation is required. If patients have not been vaccinated, they must be vaccinated at least 2 weeks prior to dosing. The choice of vaccine(s) should take into account the serotypes prevalent in the geographic areas in which study patients will be enrolled.

Exclusion Criteria:

1. Patients requiring or undergoing peritoneal dialysis.
2. Patients with a known contraindication to treatment with blood products.
3. Patients with a known pro-thrombotic disorder and/or history of thrombosis or hyper-coagulable state, excluding hemodialysis venous access clotting.
4. Patients who have positive PCR results for hepatitis B and/or hepatitis C, and/or history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
5. Patients at risk for tuberculosis (TB)
6. Patients with any severe, progressive or uncontrolled acute or chronic medical condition not related to end-stage renal disease (such as uncontrolled infectious disease or sepsis), clinical laboratory abnormalities at screening or baseline that in the investigator's opinion would make the patient inappropriate for entry into this study, or known active presence of malignancies.
7. Pregnant or nursing (lactating) women.
8. Women of child-bearing potential, unless highly effective methods of contraception are used during dosing and for 50 days after the last dose of LFG316, or sexually active males unwilling to use a condom during intercourse while taking investigational drug and for 50 days after the last dose of LFG316.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetics (PK) of LFG316: Area Under the Plasma Concentration-time Curve (AUC) | 1 month
  The following PK parameters were determined from the plasma concentration time profile of LFG316 using a non-compartmental method:
  AUClast: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
  AUCinf: Area under the plasma concentration-time curve from time zero to infinity
Plasma Pharmacokinetics (PK) of LFG316: Observed Maximum Plasma Concentration Following Drug Administration (Cmax) | 1 month

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jordan SC, Kucher K, Bagger M, Hockey HU, Wagner K, Ammerman N, Vo A. Intravenous immunoglobulin significantly reduces exposure of concomitantly administered anti-C5 monoclonal antibody tesidolumab. Am J Transplant. 2020 Sep;20(9):2581-2588. doi: 10.1111/ajt.15922. Epub 2020 May 13. PMID 32301258
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=343
- See also: Results for CLFG316B2101 can be found on Novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17183